CLINICAL TRIAL: NCT01268514
Title: ENHANCE: A Prospective Long-term EvaluatioN of the Use of Permacol™ Biological Implant in tHe Repair of Complex AbdomiNal Wall CasEs
Brief Title: ENHANCE: A Prospective EvaluatioN of Permacol™ in tHe Repair of Complex AbdomiNal Wall CasEs
Acronym: ENHANCE
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVPERH0108
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hernia, Abdominal; Abdominal Injuries
Keywords: Complex; Abdominal Wall Reconstruction; AWR; Hernia
MeSH Terms: conditions — Hernia, Abdominal; Abdominal Injuries; Hernia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this prospective study is to evaluate short-term, mid-term, and long-term clinical outcomes associated with the use of Permacol™ Biological Implant in the treatment of complex abdominal wall defects

DETAILED DESCRIPTION:
This will be a prospective, multi-centre, non-randomized study to collect post-market clinical data on Permacol™ Biological Implant following complex abdominal wall repair (including abdominal wall defects and fascial dehiscence). The subjects will have baseline and day of surgery visits performed, and then subjects will return to the investigator for evaluation of defect and safety related morbidities at follow up visits scheduled at 1 month, 6 months, 12 months, 24 months, and 36 months post-surgery.

The study will enroll up to 200 subjects at up to 20 sites. Enrollment is anticipated to take between 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will be eligible for study enrollment:

1. Subjects who are 18 years of age and older
2. Subjects of either sex
3. Subjects who require complex abdominal repair using Permacol™ Biological Implant.
4. Subjects who are willing and able to adhere to protocol requirements and provide written informed consent

Exclusion Criteria:

All subjects who meet any of the following criteria should not be enrolled into the study:

1. Subjects who are pregnant
2. Subjects with a medical condition that in the opinion of the investigator may preclude participation (e.g. Ehlers Danlos Syndrome) or interfere with completion of study follow-up
3. Subjects may not participate in any other clinical study that clinically interferes with this study while enrolled
4. Concomitant use of a synthetic or another biologic mesh
5. Subjects who require use of Permacol™ as only temporary closure with planned reoperation, or Permacol™ used as a temporary dressing in an open abdomen
6. Subject who has systemic sepsis at the time of Permacol™ implantation
7. Subject with ongoing necrotizing pancreatitis
8. Subject who requires use of Permacol™ in parastomal hernia repair alone, where there is no other anterior wall repair
9. Subject who requires prophylactic use of Permacol™ in the formation of stoma with anterior wall repair
10. Permacol™ used in pelvic floor reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who will undergo planned surgical treatment for complex abdominal wall repair with Permacol™ implantation and agree to 36 months of follow-up.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Giordano, MD, Principal Investigator — Whipps Cross University Hospital
Locations (12):
- Belgium (3):
  - AZ St Lucas, Ghent
  - CHU Ambroise Pare, Mons
  - CHU Ambroise Paré, Mons
- Universitätsklinikum des Saarlandes, Homburg, Germany
- Italy (3):
  - RCCS Istituto Clinico Humanitas di Milano, Milan
  - Istituto Nazionale Tumori, Naples
  - University Hospital (C/O Istituto Clinica Chirugica II), Rome
- Centre Hospitalier Emile Mayrisch, Esch-sur-Alzette, Luxembourg
- United Kingdom (4):
  - Whipps Cross University Hospital, Leytonstone, London
  - Royal Devon and Exeter Hospital, Exeter, Wonford
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Torbay Hospital, Torquay

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 patients were enrolled at 12 sites in 5 European countries.
Pre-assignment Details: All subjects undergoing planned surgical treatment for complex abdominal wall repair with Permacol implantation and who agree to 36 months of follow-up.
  The study allowed inclusion of up to 200 subjects at up to 20 sites.
Groups:
- Permacol Biological Implant Single Arm: Permacol Biological Implant was used to treat complex abdominal wall repairs (AWR) in this study. This was a single-arm study.
Period: Overall Study
Arm/Group | Permacol Biological Implant Single Arm
Started | 115
Participants Who Received the Device | 114
Completed | 74
Not Completed | 41
Not completed — Adverse Event | 20
Not completed — Death | 8
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 3
Not completed — Withdrawal by Surgeon | 5

BASELINE CHARACTERISTICS:
Groups:
- Permacol Biological Implant Single Arm: Permacol Biological Implant was used to treat complex abdominal wall repairs (AWR) in this study. This was a single-arm study.
  At the Screening/Baseline (-60 days) the following patient elements are collected:
  * Informed Consent
  * Demographic Information
  * Medical History
  * Surgical History
  * Concomitant Medications
  * Physical Exam
  * Radiographic Exam
Arm/Group | Permacol Biological Implant Single Arm
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 6
  Luxembourg | 22
  United Kingdom | 35
  Italy | 24
  Germany | 27
Subjects who require complex abdominal repair. [Count of Participants; unit: Participants]
  Abdominal Wall Reconstruction | 6
  Hernia | 108
Height [Mean (Standard Deviation); unit: Centimeters] | 169.0 (10.3)
Weight [Mean (Standard Deviation); unit: Kilograms] | 88.8 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hernia Recurrence or Undergo Reoperation for Hernia at 36 Months Post-surgery
Description: Characterize longitudinal outcomes at 36 months post-surgery of the proportion of subjects who undergo reoperation for hernia or hernia recurrence.
Time Frame: 36 months post-surgery
Population: This was the number of respondents at the 36-month follow up visit for this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Permacol Implant: This is the number of patients who returned for their 36 month follow-up and who were assessed for hernia recurrence.
Arm/Group | Permacol Implant
Number analyzed (Participants) | 114
Participants
  Hernia Recurrence: number analyzed (Participants) | 85
  Hernia Recurrence: Yes | 19
  Hernia Recurrence: No | 66
  Reoperation for Hernia: number analyzed (Participants) | 85
  Reoperation for Hernia: Yes | 12
  Reoperation for Hernia: No | 73

2. Secondary Outcome: Number of Participants With Short-term and Mid-term Outcomes Who Underwent Hernia Reoperation or Hernia Recurrence
Description: Characterize short-term and mid-term outcomes within 24 months post-surgery of the proportion of subjects who undergo reoperation for hernia or hernia recurrence.
Time Frame: 24 months post-surgery
Population: Proportion of subjects who underwent reoperation for hernia or hernia recurrence at 24 month post-surgery follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Permacol Biological Implant Single Arm
Number analyzed (Participants) | 91
Participants
  Patients with primary hernia requiring reoperation: Yes | 10
  Patients with primary hernia requiring reoperation: No | 61
  Patients with primary hernia requiring reoperation: Missing | 20
  Patients with hernia recurrence requiring surgery: Yes | 10
  Patients with hernia recurrence requiring surgery: No | 61
  Patients with hernia recurrence requiring surgery: Missing | 20

3. Secondary Outcome: QOL by Carolina's Comfort Scale at 6, 12, 24 and 36 Months.
Description: Quality of Life by Carolina's Comfort Scale at 6 months, 12 months, 24 months, and 36 months. The areas of assessment were: Sensation of Mesh, Pain, and Movement Limitations at each of the follow-up time points. Unscheduled surgery is any surgery that is performed outside of the primary study procedure.
  The scale measurements: 0 = no symptoms; 1 = mild but not bothersome symptoms; 2 = mild and bothersome symptoms; 3 = moderate and/or daily symptoms,;4 = severe symptoms; 5 = disabling symptoms
Time Frame: 6, 12, 24 and 36 months post-surgery. We excluded patients who were not included in this assessment at the various time-points.
Population: We excluded patients who were not included in this assessment at the 6 - 36 month post-surgery follow-up time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Permacol Implant: Permacol biological mesh implant
Arm/Group | Permacol Implant
Number analyzed (Participants) | 84
Scores on a scale
  6-month post surgery: Sensation of Mesh | 3.6 (6.0)
  6-month post surgery: Pain | 4.2 (6.9)
  6-month post surgery: Movement Limitations | 3.7 (6.3)
  12-month post surgery: Sensation of Mesh: number analyzed (Participants) | 80
  12-month post surgery: Sensation of Mesh | 3.11 (5.1)
  12-month post surgery: Pain: number analyzed (Participants) | 80
  12-month post surgery: Pain | 2.6 (4.9)
  12-month post surgery: Movement Limitations: number analyzed (Participants) | 80
  12-month post surgery: Movement Limitations | 1.9 (4.2)
  24-month post surgery: Sensation of Mesh: number analyzed (Participants) | 70
  24-month post surgery: Sensation of Mesh | 2.5 (5.5)
  24-month post surgery: Pain: number analyzed (Participants) | 70
  24-month post surgery: Pain | 2.5 (7.0)
  24-month post surgery: Movement Limitations: number analyzed (Participants) | 70
  24-month post surgery: Movement Limitations | 2.6 (6.2)
  36-month post surgery: Sensation of Mesh: number analyzed (Participants) | 65
  36-month post surgery: Sensation of Mesh | 2.6 (6.0)
  36-month post surgery: Pain: number analyzed (Participants) | 65
  36-month post surgery: Pain | 2.0 (5.6)
  36-month post surgery: Movement Limitations: number analyzed (Participants) | 65
  36-month post surgery: Movement Limitations | 2.4 (6.0)
  Unscheduled Surgery: Sensation of Mesh: number analyzed (Participants) | 3
  Unscheduled Surgery: Sensation of Mesh | 1.0 (1.7)
  Unscheduled Surgery: Pain: number analyzed (Participants) | 3
  Unscheduled Surgery: Pain | 3.0 (5.2)
  Unscheduled Surgery: Movement Limitations: number analyzed (Participants) | 3
  Unscheduled Surgery: Movement Limitations | 3.0 (5.2)

4. Secondary Outcome: Patient Satisfaction Questionnaire - Right Choice to Have Surgery
Description: Patient Satisfaction Questionnaire at 6 months, 12 months, 24 months, and 36 months.
  Question: Was it the right choice to have the surgery?
Time Frame: 6, 12, 24 and 36 months post-surgery
Population: This is the number of patients whom were included in this study assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Permacol Biological Implant Single Arm
Number analyzed (Participants) | 66
Participants
  6-month Visit: Yes | 58
  6-month Visit: No | 3
  6-month Visit: N/A | 5
  12-month Visit: number analyzed (Participants) | 65
  12-month Visit: Yes | 58
  12-month Visit: No | 1
  12-month Visit: N/A | 6
  24-month Visit: number analyzed (Participants) | 55
  24-month Visit: Yes | 46
  24-month Visit: No | 3
  24-month Visit: N/A | 6
  36-month Visit: number analyzed (Participants) | 52
  36-month Visit: Yes | 48
  36-month Visit: No | 1
  36-month Visit: N/A | 3

5. Secondary Outcome: Patient Satisfaction Questionnaire - Patient Satisfaction With Operation Outcome
Description: Patient Satisfaction Questionnaire at 6 months, 12 months, 24 months, and 36 months.
  Question: How satisfied are you with the outcome of the operation?
Time Frame: 6, 12, 24 and 36 months post-surgery
Population: This was the number of patients included in this study assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Permacol Biological Implant Single Arm
Number analyzed (Participants) | 66
Participants
  6-month: Very Satisfied | 46
  6-month: Satisfied | 16
  6-month: Somewhat Satisfied | 4
  6-month: Not Satisfied | 0
  12-month Visit: number analyzed (Participants) | 65
  12-month Visit: Very Satisfied | 45
  12-month Visit: Satisfied | 16
  12-month Visit: Somewhat Satisfied | 3
  12-month Visit: Not Satisfied | 1
  24-month Visit: number analyzed (Participants) | 55
  24-month Visit: Very Satisfied | 37
  24-month Visit: Satisfied | 13
  24-month Visit: Somewhat Satisfied | 3
  24-month Visit: Not Satisfied | 2
  36-month Visit: number analyzed (Participants) | 52
  36-month Visit: Very Satisfied | 38
  36-month Visit: Satisfied | 8
  36-month Visit: Somewhat Satisfied | 5
  36-month Visit: Not Satisfied | 1

6. Secondary Outcome: Number of Participants With Post-op Complications
Description: Subject incidence of post-operative complications, specifically: wound infection, seroma, hematoma, wound dehiscence, and fistula. Unscheduled surgery is any surgery that is performed outside of the primary study procedure.
Time Frame: 6, 12, 24 and 36 months post-surgery
Population: The overall number analyzed is the total number of patients for the study. The number analyzed in each row relates to the number of patients at each visit who had one of these adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Permacol Implant
Number analyzed (Participants) | 115
Participants
  All post-surgery visits: number analyzed (Participants) | 58
  All post-surgery visits: Wound infection | 16
  All post-surgery visits: Seroma | 18
  All post-surgery visits: Hematoma | 5
  All post-surgery visits: Wound dehiscence | 15
  All post-surgery visits: Fistula | 4
  At surgery: number analyzed (Participants) | 23
  At surgery: Wound infection | 8
  At surgery: Seroma | 3
  At surgery: Hematoma | 2
  At surgery: Wound dehiscence | 9
  At surgery: Fistula | 1
  1-month post surgery: number analyzed (Participants) | 32
  1-month post surgery: Wound infection | 7
  1-month post surgery: Seroma | 10
  1-month post surgery: Hematoma | 2
  1-month post surgery: Wound dehiscence | 12
  1-month post surgery: Fistula | 1
  6-months post surgery: number analyzed (Participants) | 16
  6-months post surgery: Wound infection | 5
  6-months post surgery: Seroma | 6
  6-months post surgery: Hematoma | 1
  6-months post surgery: Wound dehiscence | 3
  6-months post surgery: Fistula | 1
  12-months post surgery: number analyzed (Participants) | 6
  12-months post surgery: Wound infection | 1
  12-months post surgery: Seroma | 1
  12-months post surgery: Hematoma | 0
  12-months post surgery: Wound dehiscence | 1
  12-months post surgery: Fistula | 3
  24-months post surgery: number analyzed (Participants) | 0
  24-months post surgery: Wound infection | 0
  24-months post surgery: Seroma | 0
  24-months post surgery: Hematoma | 0
  24-months post surgery: Wound dehiscence | 0
  24-months post surgery: Fistula | 0
  36-months post surgery: number analyzed (Participants) | 0
  36-months post surgery: Wound infection | 0
  36-months post surgery: Seroma | 0
  36-months post surgery: Hematoma | 0
  36-months post surgery: Wound dehiscence | 0
  36-months post surgery: Fistula | 0
  Unscheduled surgeries: number analyzed (Participants) | 7
  Unscheduled surgeries: Wound infection | 2
  Unscheduled surgeries: Seroma | 2
  Unscheduled surgeries: Hematoma | 1
  Unscheduled surgeries: Wound dehiscence | 1
  Unscheduled surgeries: Fistula | 1

ADVERSE EVENTS:
Time Frame: Day of surgery, and 6, 12, 24 and 36 months post-surgery.
Arm/Group | Permacol Biological Implant Single Arm
All-Cause Mortality (participants affected / at risk) | 8/115
Serious Adverse Events (participants affected / at risk) | 93/115
Other Adverse Events (participants affected / at risk) | 41/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Permacol Biological Implant Single Arm (N=115)
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 7 (7)
Enterocutaneous Fistula (Gastrointestinal disorders) | 2 (2)
Faecal Incontinence (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2)
Intestinal Fistula (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 5 (5)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest Pain (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Allergic Granulomatous Angiitis (Immune system disorders) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1)
Device Related Sepsis (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 2 (2)
Subcutaneous Abscess (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 7 (7)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 5 (5)
Post Procedural Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1)
Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Substance-Induced Psychotic Disorder (Psychiatric disorders) | 1 (1)
Renal Failure Acute (Psychiatric disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Carotid Endarterectomy (Surgical and medical procedures) | 1 (1)
Ileostomy (Surgical and medical procedures) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Venous Thrombosis Limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Permacol Biological Implant Single Arm (N=115)
Seroma (General disorders) | 17 (18)
Recurrence of Hernia (Injury, poisoning and procedural complications) | 6 (6)
Wound Infection (Infections and infestations) | 6 (6)
Wound Dehiscence (Injury, poisoning and procedural complications) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less